CLINICAL TRIAL: NCT01667575
Title: Efficiency Study of Clarithromycin and Bismuth-containing Quadruple Therapy to Treat H.Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Dr. HONG LU, Professor of GI Division, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjkls2012004
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Functional Dyspepsia; Peptic Ulcer; Helicobacter Pylori
MeSH Terms: conditions — Peptic Ulcer | interventions — Esomeprazole; Proton Pump Inhibitors; Amoxicillin; Anti-Bacterial Agents; Clarithromycin; Bismuth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 day Quadruple Therapy (Experimental): Esomeprazole 20mg, Amoxicillin 1.0g, Clarithromycin 500mg and Bismuth Potassium Citrate 220mg,twice a day for 10 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth Potassium Citrate
- 10 day Triple therapy (Active Comparator): Esomeprazole 20mg, Amoxicillin 1.0g,and Clarithromycin 500mg, twice a day, for ten days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin
- 14 day quadruple therapy (Active Comparator): Esomeprazole 20mg, Amoxicillin 1.0g, Clarithromycin 500mg and Bismuth Potassium Citrate 220mg,twice a day for 14 days
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth Potassium Citrate; Other: long duration (14 day)

INTERVENTIONS:
Drug: Esomeprazole — antisecretary drug of the quadruple therapy
  Other Names: proton pump inhibitor
Drug: Amoxicillin — antibiotic of the quadruple therapy
  Other Names: antibiotic
Drug: Clarithromycin — antibiotic of the quadruple therapy
  Other Names: antibiotic
Drug: Bismuth Potassium Citrate — one of a component of a quadruple therapy
  Other Names: Bismuth
  Arms: 10 day Quadruple Therapy; 14 day quadruple therapy
Other: long duration (14 day)
  Arms: 14 day quadruple therapy

SUMMARY:
The purpose of this study is to observe the efficacy of ten day triple therapy-based, bismuth-containing quadruple therapy for H.pylori treatment.

DETAILED DESCRIPTION:
The success rate of currently recommended triple therapy with a proton pump inhibitor (PPI) plus amoxicillin and clarithromycin has fallen into the unacceptable range. The purpose of this study is to observe the efficacy of ten day triple therapy-based, bismuth-containing quadruple therapy for H.pylori treatment, while ten day triple therapy is used as control.

ELIGIBILITY:
Inclusion Criteria:

* patients who presented with upper gastrointestinal symptoms and endoscopically proven H.pylori-positive functional dyspepsia and scarred peptic ulcers

Exclusion Criteria:

* patients less than 18 years old, with history of H. pylori infection treatment, with previous gastric surgery, pregnancy, lactation, major systemic diseases, administration of antibiotics, bismuth, antisecretory drugs in the preceding 8 weeks, or allergy to any one of the given medication in the regimens.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | 2 months
  To calculate and compare the efficacy of 10 day and 14 day triple therapies with and without bismuth,to examine whether long duration and addition of bismuth affects the eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China